CLINICAL TRIAL: NCT00704353
Title: A Multi-Center, Randomized, Controlled Study to Investigate the Safety and Tolerability of a Single Dose of Intravenous Ferric Carboxymaltose (FCM) vs. Standard Medical Care in Treating Iron Deficiency Anemia in Subjects Who Are Not Dialysis Dependent
Brief Title: Safety and Tolerability of a Single Dose of FCM vs. Standard of Care in Treating Iron Deficiency Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1VIT08021
Record Dates: First submitted 2008-06-20; First posted 2008-06-24 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-01

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — ferric carboxymaltose; ferrous sulfate; Ferric Oxide, Saccharated; ferric gluconate; Iron-Dextran Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ferric Carboxymaltose (FCM) (Experimental): 15 mg/kg up to a maximum of 750 mg at 100 mg/minute intravenously on Day 0.
  Interventions: Drug: Ferric Carboxymaltose
- Standard Medical Care (Active Comparator): Per product label
  Interventions: Drug: Standard Medical Care (SMC)

INTERVENTIONS:
Drug: Ferric Carboxymaltose — 15 mg/kg up to a maximum of 750 mg at 100 mg/minute intravenously on Day 0.
  Arms: Ferric Carboxymaltose (FCM)
Drug: Standard Medical Care (SMC) — Per product label
  Other Names: Ferrous Sulfate, Venofer, Ferrlecit, Infed, Dexferrum
  Arms: Standard Medical Care

SUMMARY:
The objective of this study is to evaluate the safety of FCM in patients with anemia who are not dialysis dependent

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥18 years of age and able to give informed consent
* Iron deficiency is the primary etiology of anemia
* Screening Visit central laboratory Hgb indicative of anemia ≤12 g/dL
* Screening Visit ferritin indicative of iron deficiency anemia ≤100 ng/mL or ≤300 when TSAT was ≤30%

Exclusion Criteria:

* Previous participation in a FCM trial
* Known hypersensitivity reaction to FCM
* Requires dialysis for treatment of chronic kidney disease
* Current anemia not attributed to iron deficiency
* Received IV iron, RBC transfusion(s), or antibiotics 10 days prior and during the screening phase
* Anticipated need for surgery requiring general anesthesia 30 days prior to screening or during the study period
* AST of ALT greater than 1.5 times the upper limit of normal
* Received an investigational drug within 30 days of screening
* Pregnant or sexually-active females who are not able to use an effective form of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 735 (Actual)
Dates: Start 2008-06; Primary Completion 2009-07 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Luitpold Pharmaceuticals, Norristown, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospitals and medical clinics
Groups:
- Ferric Carboxymaltose (FCM): Subjects receieved an undiluted dose of iron as FCM (15mg/kg up to a maximum of 750 mg) at 100 mg/minute on Day 0.
- Standard Medical Care: Subjects received standard medical care (as determined by the Investigator) for treatment of IDA.
Period: Overall Study
Arm/Group | Ferric Carboxymaltose (FCM) | Standard Medical Care
Started | 366 | 369
Completed | 268 | 255
Not Completed | 98 | 114

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferric Carboxymaltose (FCM) | Standard Medical Care | Total
Number analyzed (Participants) | 366 | 369 | 735
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 6 | 9
  Between 18 and 65 years | 266 | 265 | 531
  >=65 years | 97 | 98 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (19.94) | 49.6 (19.88) | 49.4 (19.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 322 | 315 | 637
  Male | 44 | 54 | 98
Region of Enrollment [Number; unit: participants]
  United States | 366 | 369 | 735

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (SAE's)
Time Frame: through 30 days after the last dose of study drug (FCM or SMC for the treatment of IDA)
Measure: Number; unit: participants
Groups:
- Ferric Carboxymaltose (FCM): Subjects received an undiluted dose of iron as FCM (15 mg/kg up to a maximum of 750 mg) at 100 mg/minute on Day 0.
- Standard Medical Care: Received standard medical care (as determined by the Investigator) of IDA.
Arm/Group | Ferric Carboxymaltose (FCM) | Standard Medical Care
Number analyzed (Participants) | 366 | 369
participants | 5 | 9

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Ferric Carboxymaltose (FCM) | Standard Medical Care
Serious Adverse Events (participants affected / at risk) | 5/366 | 9/369
Other Adverse Events (participants affected / at risk) | 0/366 | 0/369
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ferric Carboxymaltose (FCM) (N=366) | Standard Medical Care (N=369)
Iron deficiency anemia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Inappropriate device stimulation of tissue (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Neuropathy (Nervous system disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less